CLINICAL TRIAL: NCT00546208
Title: Bladder Function Following Temporary Unilateral Cutaneous Ureterostomy - Long Term Follow up
Brief Title: Unilateral Cutaneous Ureterostomy - Long Term Follow up
Acronym: ureterostomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dorit Zilberman, Urology Department, Chaim Sheba Medical Center
Other Study IDs: SHEBA-07-4838-DZ-CTIL
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Bladder Function
Keywords: bladder function; cutaneous ureterostomy; hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: adolescents and young adults who underwent, as newborns, unilateral low loop cutaneous ureterostomy for severe bilateral hydro-ureteronephrosis, and that, afterwards, underwent stomal closure

SUMMARY:
This observational study is aimed at exploring bladder function following temporary unilateral low loop cutaneous ureterostomy carried out in newborns suffering from severe congenital hydro-ureteronephrosis

ELIGIBILITY:
Inclusion Criteria:

* Living patients
* Bilateral functioning kidneys
* Unilateral ureteral cutaneous diversion

Exclusion Criteria:

* Dead patients
* Single kidney
* High percutaneous ureteral diversion (e.g: cutaneous pyelostomies, bilateral cutaneous urinary diversion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adolescents and adults who had been operated in our institution for severe bilateral congenital hydro-ureteronephrosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Overall Officials: Dorit E Zilberman, MD, Principal Investigator — The Chaim Sheba Medical Center
Locations (1):
- The Chaim Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel